CLINICAL TRIAL: NCT04290507
Title: Epidemiology and Outcome of Anaphylactic Shocks Admitted to Intensive Care Unit: a French Retrospective Multicenter Study
Brief Title: Epidemiology and Outcome of Anaphylactic Shocks Admitted to Intensive Care Unit
Acronym: ANAPHYLASHOCK
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: ANAPHYLASHOCK/Guerci
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Anaphylaxis
Keywords: fluid management; mortality
MeSH Terms: conditions — Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anaphylaxis is a severe life-threatening reaction following exposure to an antigen. Its incidence is progressively increasing in the general population over years, accompanied with an increased number of hospitalizations. Although rare, this condition is often associated with a significant morbidity and mortality. The mortality rate has been recently estimated at 0.84 (95% CI, 0.79 to 0.88) per million per year in the French adult population. Age, chronic medication and cardiac or pulmonary comorbidities have been reported to increase the risk of a severe reaction. Obesity, age and cardiovascular comorbidities have been identified as risk factors for fatal anaphylaxis. However, the risk factors for death after ICU admission have not been elucidated yet.

ELIGIBILITY:
Inclusion Criteria:

* Being > 18 years old
* suffered an anaphylactic reaction, regardless of the location or causative allergen
* transferred alive in an ICU

Exclusion Criteria:

* dead within less than one hour after admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to ICU following anaphylaxis
Sampling Method: Non-Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
In-ICU mortality | Day 30
  The number of participants deceased within ICU hospitalisation

SECONDARY OUTCOMES:
Volume of fluid administered | Day 30
  The volume of fluid administered during priori to and during ICU stay, in millilitres will be noted
Amount of epinephrine | Day 30
  Quantity of epinephrine administered during ICU stay
Amount of norepinephrine | Day 30
  Quantity of norepinephrine administered during ICU stay
Number and severity of organ failure | Day 30
  The severity of organ failure will be assessed with the SOFA score
Extracorporeal life support requirement | Day 30
  The number of participants that required ECMO V/V or A/V

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital of Nancy, Nancy
  - University Hospital of Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerci P, Tacquard C, Chenard L, Millard D, Soufir L, Malinovsky JM, Garot M, Lalot JM, Besch G, Louis G, Thion LA, Charpentier C, Kimmoun A, Danguy Des Deserts M, Carreira S, Plantefeve G, Novy E, Abraham P, Mertes PM; Societe Francaise d'Anesthesie et Reanimation (SFAR) Research Network. Epidemiology and outcome of patients admitted to intensive care after anaphylaxis in France: a retrospective multicentre study. Br J Anaesth. 2020 Dec;125(6):1025-1033. doi: 10.1016/j.bja.2020.08.024. Epub 2020 Sep 12. PMID 32928517